CLINICAL TRIAL: NCT00387738
Title: A Randomized, Double-Masked, Placebo-Controlled, Multicenter, Dose-Regimen Study of the Efficacy and Safety of TOLAMBA™ in Ragweed-Allergic Rhinitis Adults
Brief Title: Efficacy and Safety Study of TOLAMBA™ in Ragweed-Allergic Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim data indicated that subjects exhibited no meaningful allergic disease during the first ragweed season, making it impossible to measure treatment effect.
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DV1-SAR-09
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Ragweed; Allergy; Allergic; Rhinitis; Hay Fever; Seasonal; Treatment; Immunotherapy; Vaccine
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity; Rhinitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): TOLAMBA™ dose-intense regimen
  Interventions: Biological: Amb a 1 immunostimulatory oligodeoxyribonucleotide conjugate
- 2 (Experimental): TOLAMBA™ lower-dose regimen
  Interventions: Biological: Amb a 1 immunostimulatory oligodeoxyribonucleotide conjugate
- 3 (Placebo Comparator)
  Interventions: Biological: Histamine base

INTERVENTIONS:
Biological: Amb a 1 immunostimulatory oligodeoxyribonucleotide conjugate — Escalating doses, 6 weekly subcutaneous (under the skin) injections
  Other Names: TOLAMBA™
  Arms: 1; 2
Biological: Histamine base — Escalating doses, 6 weekly subcutaneous (under the skin) injections
  Arms: 3

SUMMARY:
The purpose of this study is to find out if a new investigational vaccine, TOLAMBA™, is safe and effective in reducing the symptoms of ragweed allergy.

DETAILED DESCRIPTION:
Ragweed allergy is the most common seasonal allergy in North America. Allergen immunotherapy is a therapeutic option for patients who have allergy symptoms that cannot be adequately controlled by avoidance of the allergen or medication. It may also be appropriate for those who cannot tolerate their medications due to side effects or have difficulties with medication compliance. This study compares the safety and efficacy of two different dosing regimens of TOLAMBA™ with placebo in reducing the symptoms of ragweed-allergic adults over two consecutive ragweed pollen seasons.

Comparison(s): Subject-rated allergy symptoms of subjects treated with TOLAMBA™ dose-intense regimen or TOLAMBA™ lower-dose regimen, compared with subjects treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Has a history of ragweed allergic rhinitis (hayfever) during at least the last 2 consecutive seasons that has required treatment with antihistamines, decongestants and/or nasal steroids, but where symptom relief has been incomplete
* Is willing to stay in their ragweed area during the historical peak period of the local ragweed season, and willing to travel for no more than 2 weeks (cumulative time) outside of their ragweed area during the entire season

Exclusion Criteria:

* Has had any hospital admissions for asthma
* Has smoked within the past year, or has a ≥10-pack per year smoking history
* Has had any previous immunotherapy with ragweed pollen extract, or was in a previous clinical trial with TOLAMBA™
* Has used Xolair within the past 12 months
* Has a history of anaphylaxis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 738 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total nasal symptom score during the peak period of the ragweed pollen season. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martins, MD, DPhil, Study Director — Dynavax Technologies Corporation
Locations (28):
- United States (28):
  - Center Of Research Excellence, Oxford, Alabama
  - Atlanta Allergy & Asthma Clinic, Stockbridge, Georgia
  - Clinical Research of Atlanta, Stockbridge, Georgia
  - Sneeze, Wheeze, and Itch Associates, Normal, Illinois
  - Research Center of Indiana, Indianapolis, Indiana
  - Asthma and Allergy Research Center, Minneapolis, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - Clinical Research of the Ozarks, Columbia, Missouri
  - Clinical Research of The Ozarks, Rolla, Missouri
  - Clinical Research Center, St Louis, Missouri
  - Clinical Research of the Ozarks, Warrensburg, Missouri
  - Midwest Allergy & Asthma Clinic, Omaha, Nebraska
  - Creighton University, Omaha, Nebraska
  - Asthma & Allergy Center, Papillion, Nebraska
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Allergy & Asthma Center, High Point, North Carolina
  - Allergy & Respiratory Center, Canton, Ohio
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Asthma & Allergy Research Associates, Upland, Pennsylvania
  - AARA Research Center, Dallas, Texas
  - Pharmaceutical Research & Consulting, Dallas, Texas
  - Kerrville Allergy and Asthma Associates, Kerrville, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research, San Antonio, Texas
  - Asthma, Allergy & Sinus Center, Greenfield, Wisconsin
  - University of Wisconsin Madison Medical School, Madison, Wisconsin
  - Advanced Healthcare, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
The IND for Tolamba was withdrawn, it was reported to the agency that there was no plan to conduct clinical studies with this compound. [per email from EA 18Dec2015. 3/1/2017 - No update

REFERENCES:
- See also: American Academy of Allergy, Asthma & Immunology — http://www.aaaai.org
- See also: Dynavax Web Page — http://www.dynavax.com